CLINICAL TRIAL: NCT04884412
Title: Deep Brain Stimulation for Parkinson's Disease: Probabilistic STN Targeting Under General Anaesthesia Without Micro-electrode Recordings (MER) vs Current Targeting Procedure
Brief Title: Deep Brain Stimulation for Parkinson's Disease: Probabilistic STN Targeting Under General Anaesthesia Without Micro-electrode Recordings vs Current Targeting Procedure
Acronym: PARKEO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2019/54
Record Dates: First submitted 2021-04-27; First posted 2021-05-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Deep brain stimulation; Sub-thalamic nucleus; Parkinson Disease; Micro-electrode recordings; DBS targeting
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: National multicentre, prospective, randomised, non-inferiority, open label, comparative clinical trial in 2 parallel groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PARKEO 2 targeting with asleep deep brain stimulation procedure (Experimental): Participant with parkeo 2 targeting procedure
  Interventions: Procedure: Surgery under general anesthesia with experimental targeting
- Usual DBS procedure (Active Comparator): Participant with usual targeting and surgery
  Interventions: Procedure: Usual Surgery

INTERVENTIONS:
Procedure: Surgery under general anesthesia with experimental targeting — Surgery will be performed under general anesthesia. The electrodes will be inserted directly on the targets without MER, with PARKEO_2 targets provided by the Bordeaux University Hospital, based on the machine-learning model developed in Bordeaux.
  Arms: PARKEO 2 targeting with asleep deep brain stimulation procedure
Procedure: Usual Surgery — In the control group, surgery will be performed as usual in each centre under local or general anaesthesia. This group represents the current state of the art of deep brain stimulation in these centres.
  Arms: Usual DBS procedure

SUMMARY:
Deep brain stimulation (DBS) of the sub-thalamic nucleus (STN) has evolved over the past decades as a mainstream therapy for advanced Parkinson's disease (PD). The classical procedure consists in STN indirect targeting based on stereotactic atlases or statistical coordinates in AC-PC (Anterior Commissure - Posterior Commissure) referential along with target control and correction by micro-electrode recordings (MER) and awake clinical testing. To avoid potential complications and patient discomfort related to current procedure, asleep surgery without this control process has become more and more performed, essentially thanks to the progress of neuroimaging allowing to STN visualization. However, it has been reported a relative inaccuracy between the "radiological" STN delimitated on several types of MRI sequences (T2, T2*, SWI) and the per-operative electrophysiological findings. As a result, there are currently many types of STN-DBS procedures, and the lack of standardization between techniques complicates the interpretation of postoperative results on anatomical, electrophysiological and clinical points of view. Furthermore, to date, it has not been proven that asleep surgery without MER and clinical controls is as effective as the standard procedure in a prospective controlled randomized clinical trial.

Investigators hypothesize that the clinical-based 18 landmarks STN target will be precise enough to allow to perform surgery under general anesthesia without MER correction, and accurate enough to achieve non inferior clinical results compared to what is usually done in each centre.

The main objective is to compare at one year, the % of motor improvement after PARKEO 2-targeting asleep DBS without intraoperative MER versus the targeting procedure using intraoperative MER by the UPRDRS 3 (Unified Parkinson's disease rating scale 3).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of idiopathic Parkinson's disease at the stage of motor fluctuations despite optimal medical treatment
* L-DOPA sensitivity defined by motor improvement above 50% on the UPDRS-3 scale after a dose of 150% of the usual early morning treatment
* Indication for STN-DBS approved by the local multidisciplinary movement disorders committee.
* Patients between 18 and 70 years of age
* Patients covered by a health insurance scheme
* Signed informed consent.

Exclusion Criteria:

* Significant cognitive decline defined as a score < 22 on the MoCA scale
* Mood disorders defined by a score > 20 on the Beck Depression Inventory
* Significant cortical atrophy or leukoencephalopathy visualised by brain MRI
* Contraindication to anaesthesia and MRI
* Lack of contraceptive treatment for women with ability to procreate
* Pregnant or breast-feeding woman
* Unstoppable anticoagulant or antiaggregant treatment
* Persons under legal protection (Persons deprived of liberty or incapable of giving consent or under curatorship or tutorship…)
* Patient with severe psychiatric disorders (on Diagnostic and Statistical Manual of Mental Disorders IV)
* Inability to follow the patient until the end of study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Stimulation efficacy | 12 months after surgery (M12)
  The primary endpoint is the efficacy of the stimulation on motor symptoms assessed by the change in UPDRS-3 scores between OFF and ON stimulation evaluations at one year after surgery without any medical treatment (OFF medication).
  Unified Parkinson's Disease Rating Scale 3 (UPDRS 3) questionnaire: 0 to 132 points, with the highest score indicating worsening

SECONDARY OUTCOMES:
Quality of life assessment | inclusion (Month-1) and 12 months after surgery (M12)
  Quality of life on the Parkinson Disease Questionnaire 39 (PDQ39) scale assessed by the change in PDQ39 scores.
  PDQ 39 questionnaire : 0 to 156 points, with the highest score indicating worsening condition
Stereotactic accuracy | Surgery intervention (Month 0)
  Stereotactic accuracy as measured by the Euclidian distance between active contact location and intra-operative defined target in each group
Operative characteristics (1) | Surgery intervention (Month 0)
  Operative characteristic : procedure length
Operative characteristics (2) | Surgery intervention (Month 0)
  Operative characteristic : radiation dose
Operative characteristics (3) | Surgery intervention (Month 0)
  Operative characteristic : pneumocephalus
Operative characteristics (4) | Surgery intervention (Month 0)
  Operative characteristic : and length of hospital stay (in days).
Distance between active contact location and preoperative target | Surgery intervention (Month 0)
  Distance between active contact location and preoperative defined target in each group
Improvement of UPDRS3 | 12 months after surgery (M12)
  The percentage of improvement of UPDRS3 calculated between the preoperative OFF and the post-operative ON stimulation scores at one year and compared between the two groups.
  Unified Parkinson's Disease Rating Scale 3 (UPDRS 3) questionnaire: 0 to 132 points, with the highest score indicating worsening
Efficacy of the targeting procedure on motor symptoms (1) | 12 months after surgery (M12)
  The efficacy of the targeting procedure on motor symptoms assessed by the change in UPDRS-3 scores between OFF and ON stimulation evaluations at one year after surgery without any medical treatment (OFF medication). The change will be calculated as a difference between the OFF and ON stimulation scores at one year.
  Unified Parkinson's Disease Rating Scale 3 (UPDRS 3) questionnaire: 0 to 132 points, with the highest score indicating worsening
Efficacy of the targeting procedure on motor symptoms (2) | 12 months after surgery (M12)
  The efficacy of the targeting procedure on motor symptoms compared to the efficacy of L-DOPA by the change in UPDRS-3 scores between OFF and ON stimulation evaluations at one year after surgery without any medical treatment (OFF medication). The change will be calculated as a ratio between the effect of stimulation alone versus medication alone at one year.
  Unified Parkinson's Disease Rating Scale 3 (UPDRS 3) questionnaire: 0 to 132 points, with the highest score indicating worsening
reduction in the levodopa equivalent daily doses (LEDD) | 12 months after surgery (M12)
  The reduction in the levodopa equivalent daily doses (LEDD) from the baseline and one year (a 100-mg daily dose of standard levodopa is equivalent to the following doses of other medications: 133 mg of controlled-release levodopa; 75 mg of levodopa plus entacapone; 1 mg of pergolide, pramipexole lisuride, or cabergoline; 5 mg of ropinirole; 10 mg of bromocriptine or apomorphine; and 20 mg of dihydroergocryptine) will be evaluated
Post-operative cognitive | 12 months after surgery (M12)
  Post-operative cognitive will be assess by the difference from the baseline and one year using MDRS.
  Mattis Dementia Rating Scale: 0 to 144 points, with the most important score indicating improvement in condition
Post-operative mood | 12 months after surgery (M12)
  Post-operative mood will be assess by the difference from the baseline and one year using BDI scale.
  Beck Depression Inventory (BDI): 0 to 63 points, with the most important score indicating worsening condition
Intra and post-operative surgical complications | Surgery intervention (Month 0)
  Intra and post-operative surgical complications (haemorrhage, infection, neuromodulation-related side effects) will be prospectively collected and assessed
Total cost of each procedure (PARKEO-2 targeting compared to targeting procedure using intraoperative MER) | Surgery intervention (Month 0)
  A cost analysis will be performed to assess all hospital resources
Cost-effectiveness ratio, expressed in terms of cost per Qaly gained at 1 year | 12 months after surgery (M12)
  This ratio will provide useful information about the costs (avoided or additional) required to gain a Qaly, one year after surgery, from the French healthcare system point of view

CONTACTS AND LOCATIONS:
Overall Officials: Julien ENGELHARDT, Dr, Principal Investigator — University Hospital, Bordeaux; Emmanuel CUNY, Pr, Study Director — University Hospital, Bordeaux; Antoine BENARD, Dr, Study Chair — University Hospital, Bordeaux
Locations (8):
- France (8):
  - CHU Amiens, Amiens
  - CHU de Bordeaux, Bordeaux
  - Hospices Civils de Lyon, Lyon
  - CHU Marseille, Marseille
  - CHU de Nice, Nice
  - CHU de Rouen, Rouen
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse